CLINICAL TRIAL: NCT05310149
Title: Measuring the Influence of Maxillary Obturator Prosthesis on Facial Morphology in Patient With Unilateral Maxillary Defects Using Stereophotogrammetry
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hoor Nafae, Master Degree Candidate, Cairo University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7122
Record Dates: First submitted 2022-03-25; First posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Facial Asymmetry
MeSH Terms: conditions — Facial Asymmetry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- obturator group(unilalateral maxillary defect) (Experimental): Prosthetic intervention with maxillary obturator prosthesis is necessary to restore the contours of the resected palate and to recreate the functional separation of the oral cavity and sinus and nasal cavities. Followings are the objectives of maxillary obturator Restoration of esthetics or cosmetic appearance of the patient, Restoration of function, Protection of tissues, Therapeutic or healing effect and psychological therapy.
  Interventions: Device: Prosthetic intervention with maxillary obturator prosthesis
- Control group (No Intervention): intact side of the same patient

INTERVENTIONS:
Device: Prosthetic intervention with maxillary obturator prosthesis — Prosthetic intervention with maxillary obturator prosthesis is necessary to restore the contours of the resected palate and to recreate the functional separation of the oral cavity and sinus and nasal cavities. Followings are the objectives of maxillary obturator Restoration of esthetics or cosmetic appearance of the patient, Restoration of function, Protection of tissues, Therapeutic or healing effect and psychological therapy.
  Arms: obturator group(unilalateral maxillary defect)

SUMMARY:
Functional rehabilitation and quality of life after maxillofacial surgery have been emphasized in recent years. It depends mainly on outcomes of maxillofacial reconstruction and rehabilitation involving functions, esthetics, psychology acceptance and resocialization.

Tooth loss, alveolar and maxillary bone resorption or changes of the hard palate cause facial asymmetry in patient with maxillofacial surgery. The facial soft tissue over the defect become recessed as a result of loss of lip and buccal support which lead to decrease the quality of life and psychological disorders. Prosthetic intervention with maxillary obturator prosthesis is necessary to restore the contours of the resected palate and to recreate the functional separation of the oral cavity and sinus and nasal cavities. The purpose of this study is to investigate the influence of maxillary obturator on facial morphology in patient with unilateral maxillary defect by using 3 dimensional digital stereophotogrammetry compared to the intact side of the same patient

ELIGIBILITY:
Inclusion Criteria:

* adult patient of both sexes, 6 months after partial maxillectomy with good periodontal condition of remaining tooth especially abutment tooth.

Exclusion Criteria:

* patient with history of radiotherapy, bad oral hygiene patient with tumor recurrence, patient with mental instability, patient with systemic disorders like uncontrolled diabetes, compromised heart function

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2022-01-07 (Actual); Primary Completion 2022-10-15 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Facial morphology | after 6 months of maxillofacial surgery
  3 dimensional digital stereophotogrammetry compared to the intact side of the same patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Hoor Nafade, Zagazig, Egypt